CLINICAL TRIAL: NCT05332028
Title: Comparison of the Analgesic Efficacy of Ultrasound-guided Paravertebral Block and Mid-point Transverse Process Pleura Block in Mastectomy Surgery
Brief Title: Ultrasound-guided Paravertebral Block Versus Mid-point Transverse Process Pleura Block in Mastectomy Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet AKSOY, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/1/6
Record Dates: First submitted 2022-04-02; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Mastectomy; Lymphedema; Anesthesia, Local; Surgery
Keywords: mastectomy; anesthesia; paravertebral block; mid-Point Transverse Process Pleura block; patient-controlled analgesia
MeSH Terms: conditions — Lymphedema | interventions — Bupivacaine; Needles; Propofol; Fentanyl

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to Group 1 (Patients undergoing PVB) or Group 2 (Patients undergoing MTP block) for a ratio of 1:1, including 32 patients each, using a computer-generated table of random numbers and concealed sealed opaque envelopes. An investigator opened the sealed opaque envelopes before the block application.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study was planned as triple-blind; patients and investigators were blinded to the group allocation. An investigator opened the sealed opaque envelopes before the block application. An another anaesthetist who was blinded to the group assignment was responsible for collecting intra-and postoperative data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Patients undergoing paravertebral block (Experimental): After cleaning the area with antiseptic solution, the sterilized linear USG probe (Esaote MyLab30®, CA631 high-frequency probe, United Kingdom) was covered. The flat probe was placed between two transverse processes on the paramedian plane; transverse processes, superior costotransverse ligament and pleura were consecutively visualized. The linear ultrasound probe was fixed to the T3-T4 vertebra level. The skin and subcutaneous tissue were anaesthetized with 2% lidocaine, then 22 gauge 100 mm needle (Stimuplex ®; B Braun, Melsungen, Germany) was led in a cranial-cephalic direction to the paravertebral gap. Trapezius, rhomboid, erector spinae muscles were crossed by seeing the tip of the needle. Transverse processes were reached and the intercostal muscles were passed. When the needle reached the paravertebral level, a 20 mL of 0.25% bupivacaine was applied as a single administration.
  Interventions: Drug: bupivacaine; Device: 22 gauge 100 mm needle; Drug: Propofol; Drug: fentanyl
- Group 2: Patients undergoing Mid-Point Transverse Process Pleura (MTP) block (Active Comparator): After cleaning the area with antiseptic solution, the sterilized linear USG probe (Esaote MyLab30®, CA631 high-frequency probe, United Kingdom) was covered. The flat probe was placed between two transverse processes on the paramedian plane; transverse processes, superior costotransverse ligament and pleura were consecutively visualized. The linear ultrasound probe was fixed to the T3-T4 vertebra level. The skin and subcutaneous tissue were anaesthetized with 2% lidocaine, then 22 gauge 100 mm needle (Stimuplex ®; B Braun, Melsungen, Germany) was led in a cranial-cephalic direction to the paravertebral gap. Trapezius, rhomboid, erector spinae muscles were crossed by seeing the tip of the needle. Transverse processes were reached and the intercostal muscles were passed. When the needle reached the midpoint level between the transverse process and pleura, a 20 mL of 0.25% bupivacaine was applied as a single administration.
  Interventions: Drug: bupivacaine; Device: 22 gauge 100 mm needle; Drug: Propofol; Drug: fentanyl

INTERVENTIONS:
Drug: bupivacaine — Block applications
Device: 22 gauge 100 mm needle — Block applications
  Other Names: needle
Drug: Propofol — Routine general anesthesia protocol
Drug: fentanyl — patient-controlled analgesia

SUMMARY:
This study was performed to analyze the postoperative analgesic effects of the paravertebral block (PVB) and Mid-Point Transverse Process Pleura (MTP) block after a unilateral mastectomy surgery.

This study included 64 women aged 18-65 years, American Society of Anesthesiologists score I-III, who were scheduled for unilateral simple mastectomy operation due to breast cancer. Patients were randomly assigned to Group 1 (Patients undergoing PVB) or Group 2 (Patients undergoing MTP block) for a ratio of 1:1, including 32 patients each, using a computer-generated table of random numbers and concealed sealed opaque envelopes.

Patients were placed in the prone position. The linear ultrasound probe was fixed to the T3-T4 vertebra level. The skin and subcutaneous tissue were anaesthetized with 2% lidocaine, then 22 gauge 100 mm needle was led in a cranial-cephalic direction to the paravertebral gap. Trapezius, rhomboid, erector spinae muscles were crossed by seeing the tip of the needle. Transverse processes were reached and the intercostal muscles were passed. When the needle reached the paravertebral level in Group 1, and the midpoint level between the transverse process and pleura in Group 2, it was observed that there was no blood or air by aspiration. Then, the needle location was confirmed with 0.5-1 mL of saline, and a 20 mL of 0.25% bupivacaine was applied. Thirty minutes after block application, the sensorial block level was evaluated by pinprick test at the midclavicular line, and the blocked dermatome area was recorded as front and back. Complications developed during the process (such as hypotension, vascular injury, local anaesthetic toxicity) were recorded.Routine general anesthesia protocol was performed to all patients.At the end of the surgery, neuromuscular block antagonization was performed with 4 mg/kg sugammadex. All of the patients were extubated and taken to the postanesthetic care unit (PACU). In the PACU, a patient-controlled analgesia device (PCA) containing fentanyl was administered.

Time to the first request for analgesia, postoperative fentanyl consumption, and VAS score values at rest and in motion at postoperative 1, 4, 8, 12, 16, 20 and 24 hours, the duration of block implementation and the duration of surgery were recorded.

DETAILED DESCRIPTION:
This prospective randomized controlled trial was performed to analyze the postoperative analgesic effects of the paravertebral block (PVB) and Mid-Point Transverse Process Pleura (MTP) block after a unilateral mastectomy surgery.

This prospective randomized placebo-controlled triple-blind study was approved by the Ethical Committee of Ataturk University, Medical Faculty, Erzurum, Turkey. The study was carried out at the Anesthesiology and Reanimation Department of Ataturk University, Medical Faculty, Erzurum, Turkey.This study included 64 women aged 18-65 years, American Society of Anesthesiologists score I-III, who were scheduled for unilateral simple mastectomy operation due to breast cancer.The day before surgery, patients were assessed by a researcher who was blind to group assignment. All patients were informed about the study, and written informed consent was obtained from all participants who agreed to participate in the study.

This study was planned as triple-blind; patients and investigators were blinded to the group allocation. The patients were fasted for 8 hours before surgery. Before the anesthesia procedure, demographic data of all patients (age, weight, height, ASA physical status), baseline values of heart rate, systolic, diastolic and average blood pressure were recorded. Vascular access was established for all patients via 22-gauge intravenous cannula, and premedication was provided using 0.03 mg/kg of IV midazolam. Patients were randomly assigned to Group 1 (Patients undergoing PVB) or Group 2 (Patients undergoing MTP block) for a ratio of 1:1, including 32 patients each, using a computer-generated table of random numbers and concealed sealed opaque envelopes. An investigator opened the sealed opaque envelopes before the block application. An another anesthetist who was blinded to the group assignment was responsible for collecting intra-and postoperative data. All surgeries were done by the same surgical and anaesthetic teams.

All blocks were fulfilled by the same anesthesiologist, who had at least five years of experience in the profession, with the help of a flat probe (1-8 MHz) and using 22 gauge, 100 mm insulated facet tip needles before general anesthesia. Patients were placed in a sitting position, spinous processes were marked starting from the C7 spinous process to the T6 level. Then, patients were placed in the prone position. After cleaning the area with antiseptic solution, the sterilized linear ultrasonography probe (Esaote MyLab30®, CA631 high-frequency probe, United Kingdom) was covered. The flat probe was placed between two transverse processes on the paramedian plane; transverse processes, superior costotransverse ligament and pleura were consecutively visualized. The linear ultrasound probe was fixed to the T3-T4 vertebra level. The skin and subcutaneous tissue were anesthetized with 2% lidocaine, then 22 gauge 100 mm needle (Stimuplex ®; B Braun, Melsungen, Germany) was led in a cranial-cephalic direction to the paravertebral gap. Trapezius, rhomboid, erector spinae muscles were crossed by seeing the tip of the needle. Transverse processes were reached and the intercostal muscles were passed. When the needle reached the paravertebral level in Group 1, and the midpoint level between the transverse process and pleura in Group 2, it was observed that there was no blood or air by aspiration. Then, the needle location was confirmed with 0.5-1 mL of saline, and a 20 mL of 0.25% bupivacaine was applied. Local anesthetic dissemination was seen in both cranial and caudal directions. Thirty minutes after block application, the sensorial block level was evaluated by pinprick test (normal sensation:0, decreased sensation:1, insensitivity:2) at the midclavicular line, and the blocked dermatome area was recorded as front and back. The duration from placing the patient in the prone position to removing the needle used for the block procedure was defined as the block application duration and recorded. Complications developed during the process (such as hypotension, vascular injury, local anesthetic toxicity) were recorded.

Routine general anesthesia protocol was performed using 2-3 mg/kg IV propofol, 2 µg/kg IV fentanyl and 0.6 mg/kg IV rocuronium. Anesthesia was maintained with desflurane, a fresh gas flow of 3 L/min and a nitrous oxide mixed with oxygen in a 2:1 ratio. During surgery, the patients' systolic, diastolic and average artery blood pressures and oxygen saturation values were recorded in the 5th, 10th, 15th, 20th, 35th, and 50th minutes, and postoperative 1st and 2nd hours. All operations were performed by the same surgical team using the same surgical technique.

At the end of the surgery, neuromuscular block antagonization was performed with 4 mg/kg sugammadex. All of the patients were extubated and taken to the postanesthetic care unit (PACU). Patients with a modified Aldrete score of 9 and above were transferred to the clinic. At the end of the surgery, IV 1g of paracetamol was administered to all patients. The same dose was repeated every 6 hours postoperatively. To prevent postoperative nausea and vomiting, IV 8 mg of ondansetron was administered to all patients. Intravenous ephedrine (6 mg) was used to treat hypotension (a 20% decrease in systolic blood pressure compared to preoperative values) and IV atropine (1 mg) was given in case of bradycardia (the heart rate < 45 beats/minute) during surgery. When nausea and vomiting were observed, intravenous metoclopramide (10 mg) was administered.

In the PACU, a patient-controlled analgesia device (PCA) containing fentanyl was administered. The PCA was set at a 10 μg/mL concentration, with a 50 μg loading dose, 10 minutes lockout duration, a bolus of 25 μg, and without basal infusion, and it was left connected for 24 hours. Postoperative fentanyl consumption was recorded as 0-4 hours, 4-8 hours, 8-12 hours, 12-16 hours, 16-20 hours, 20-24 hours and 24 hours total. A patient-controlled analgesia device (PCA), which contains fentanyl at a concentration of 10 mcg/ml, with a loading dose of 50mcg, a lock-out duration of 10 minutes, a bolus dose of 25 mcg, and no basal infusion, was connected to all patients in the PACU. Postoperative pain was assessed using Visual Analog Pain Scale (VAS), which ranged from 0 (no pain) to 10 (worst imaginable pain) in the postoperative 1, 4, 8, 12, 16, 20 and 24th hours. Patients with a VAS score of 4 and above received 25 mg of rescue meperidine. The incidence of nausea and vomiting was recorded in the postoperative first 24 hours. Postoperative follow-up of the cases was done by an independent observer who was blinded to the group assignment.

Time to the first request for analgesia, postoperative fentanyl consumption, and VAS score values at rest and in motion at postoperative 1, 4, 8, 12, 16, 20 and 24 hours, the duration of block implementation and the duration of surgery were recorded.

Power analysis for the study was calculated using the NCSS-PASS (NCSS LLC, Kaysville, Utah) software. The primary end point of the study was the total opioid consumption for the first 24 hours postoperatively. The minimum sample size required for this study was calculated based on Gürkan et al.'s study. They reported that the difference between groups opioid requirements in the first 24 hours after surgery was 1.5; the common standard deviation within a group was assumed to be 3.43 and 4.15. As a result of a power analysis, the sample size for a group was determined to be 30 patients with a power of 80% and alpha of 5%. It was planned to include 64 patients throughout the study, 32 patients in each group, considering potential dropouts.

The SPSS 20 package software was used for data analysis. Numerical data were expressed as mean and standard deviation, categorical data were presented as numbers (n) and percentages (%). The normal distribution of data were evaluated using a the Kolmogorov-Smirnov Z test. Independent sample t-test was used for the analysis of parametric data and Mann-Whitney U test was used for the analysis of non-parametric data. Analysis of repetitive measurements in intra-group comparisons was done with ANOVA, analysis of categorical data was done using chi-square test. The results were considered statistically significant if p value<0.05.

ELIGIBILITY:
Inclusion Criteria:

* All patients were informed about the study, and written informed consent was obtained from all participants who agreed to participate in the study.
* aged 18-65 years
* ASA I-III
* scheduled for unilateral simple mastectomy operation due to breast cancer.

Exclusion Criteria:

* ASA >3
* BMI≥35
* bleeding diathesis
* neurological disease
* infections at the needle site
* a history of allergy to any of the drugs used in the study
* those who had undergone axillary lymph dissection

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — who were scheduled for unilateral simple mastectomy operation due to breast cancer.
Enrollment: 64 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
to compare the postoperative opioid consumption in the first 24 hours after surgery | Fentanyl consumption in the postoperative 24 hours.
  All of the patients were extubated and taken to the postaesthetic care unit (PACU).In the PACU, a patient-controlled analgesia device (PCA) containing fentanyl was administered.

SECONDARY OUTCOMES:
to compare postoperative pain scores at rest and in motion. | The first 24 hours after surgery.
  Postoperative pain was assessed using VAS, which ranged from 0 (no pain) to 10 (worst imaginable pain).
time to the first opioid analgesic request. | immediately after the surgery.
  Postoperative follow-up of the cases was done by an independent observer.
the amount of rescue analgesics | The first 24 hours after surgery.
  Patients with a VAS score of 4 and above received rescue analgesic.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur DOSTBIL, Study Director — Department of Anesthesiology and Reanimation; Ilker INCE, Principal Investigator — Department of Anesthesiology and Reanimation; Erdem KARANENIZ, Principal Investigator — Department of General Surgery
Locations (1):
- Mehmet Aksoy, Erzurum, string:Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
participants do not allow data to be shared.

REFERENCES:
- [Background] Waks AG, Winer EP. Breast Cancer Treatment: A Review. JAMA. 2019 Jan 22;321(3):288-300. doi: 10.1001/jama.2018.19323. PMID 30667505
- [Background] Loibl S, Poortmans P, Morrow M, Denkert C, Curigliano G. Breast cancer. Lancet. 2021 May 8;397(10286):1750-1769. doi: 10.1016/S0140-6736(20)32381-3. Epub 2021 Apr 1. PMID 33812473
- [Background] Fecho K, Miller NR, Merritt SA, Klauber-Demore N, Hultman CS, Blau WS. Acute and persistent postoperative pain after breast surgery. Pain Med. 2009 May-Jun;10(4):708-15. doi: 10.1111/j.1526-4637.2009.00611.x. Epub 2009 Apr 22. PMID 19453965
- [Background] Lam S, Qu H, Hannum M, Tan KS, Afonso A, Tokita HK, McCormick PJ. Trends in Peripheral Nerve Block Usage in Mastectomy and Lumpectomy: Analysis of a National Database From 2010 to 2018. Anesth Analg. 2021 Jul 1;133(1):32-40. doi: 10.1213/ANE.0000000000005368. PMID 33481402
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH. Erector spinae plane block and thoracic paravertebral block for breast surgery compared to IV-morphine: A randomized controlled trial. J Clin Anesth. 2020 Feb;59:84-88. doi: 10.1016/j.jclinane.2019.06.036. Epub 2019 Jul 4. PMID 31280100
- [Result] Ghoncheh M, Pournamdar Z, Salehiniya H. Incidence and Mortality and Epidemiology of Breast Cancer in the World. Asian Pac J Cancer Prev. 2016;17(S3):43-6. doi: 10.7314/apjcp.2016.17.s3.43. PMID 27165206
- [Result] DeSantis CE, Bray F, Ferlay J, Lortet-Tieulent J, Anderson BO, Jemal A. International Variation in Female Breast Cancer Incidence and Mortality Rates. Cancer Epidemiol Biomarkers Prev. 2015 Oct;24(10):1495-506. doi: 10.1158/1055-9965.EPI-15-0535. Epub 2015 Sep 10. PMID 26359465
- [Derived] Kahramanlar AA, Aksoy M, Ince I, Dostbil A, Karadeniz E. The Comparison of Postoperative Analgesic Efficacy of Ultrasound-Guided Paravertebral Block and Mid-Point Transverse Process Pleura Block in Mastectomy Surgeries: A Randomized Study. J Invest Surg. 2022 Sep;35(9):1694-1699. doi: 10.1080/08941939.2022.2098544. Epub 2022 Jul 17. PMID 35848451